CLINICAL TRIAL: NCT01367886
Title: Comparative Urine Proteomic Studies of Overactive Bladder in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: WS473527
Record Dates: First submitted 2011-05-19; First posted 2011-06-07 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Overactive Bladder
Keywords: Urine proteomics; overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fesoterodine (Other): Females with overactive bladder symptoms will be given Fesoterodine 4 mg. daily for six weeks.
  Interventions: Drug: fesoterodine

INTERVENTIONS:
Drug: fesoterodine — Fesoterodine 4 mg. tablet by mouth daily for six weeks
  Other Names: Toviaz

SUMMARY:
This study is being done to evaluate the use of a new technology (urine proteomics) - the study of proteins in the urine to identify urine markers of overactive bladder (OAB) from a simple voided urine specimen.

DETAILED DESCRIPTION:
The objectives of the study are:

1. to improve the diagnosis of overactive bladder using a non-invasive technology (urine proteomics) and
2. to study how potential urine biomarkers changes with overactive bladder symptoms after patients have been treated with fesoterodine, an FDA approved drug for the treatment of overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

For healthy volunteers the inclusion criteria are:

1. Females ≥ 18 years old
2. Not experiencing overactive bladder symptoms
3. Not experiencing frequency or urgency

For overactive bladder patients the inclusion criteria are

1. Females ≥ 18 years old
2. Overactive bladder symptoms for ≥ 3 months before screening ) Recurrent urinary tract infections (UTIS) > 3/year

Exclusion Criteria:

For healthy volunteers the exclusion criteria are:

1. Overactive bladder symptoms, such as frequency and urgency
2. Intermittent/unstable use of bladder medications
3. Pregnant women or women unwilling to use contraceptives
4. Neurological conditions: stroke, Multiple Sclerosis (MS), Parkinson's, spinal cord injury
5. Significant pelvic organ prolapsed (grade 3 or above based on physical exam)
6. Lower urinary tract surgery within past 6 months
7. Known history of IC or pain associated with OAB
8. Urinary retention requiring catheterization, indwelling catheter of Self-cath
9. Recurrent UTIS > 3/year

For overactive bladder patients the exclusion criteria are:

1. Contraindications to Fesoterodine use such as hypersensitivity, GI and urinary retention, and Glaucoma
2. Intermittent/unstable use of bladder medications
3. Pregnant women or women unwilling to use contraceptives
4. Neurological conditions: stroke, MS, Parkinson's, spinal cord injury
5. Significant pelvic organ prolapsed (grade 3 or above based on physical exam)
6. Lower urinary tract surgery within past 6 months
7. Known history of Interstitial Cystitis (IC) or pain associated with OAB
8. Urinary retention requiring catheterization, indwelling catheter of Self-cath
9. Recurrent urinary tract infections (UTIS) > 3/year

Deferral Criteria:

Treatment with OAB medications within 2 weeks before baseline visit. If patient is currently on OAB medications the patient will be asked to stop OAB medication for 2 weeks and return for baseline visit.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Henry Lai, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with overactive bladder were recruited from principal investigator's clinic practice.
Pre-assignment Details: Overactive bladder subjects completed a 3-day bladder diary and the Overactive Bladder questionnaire (OAB-q) prior to starting Toviaz (Fesoterodine) 4 mg daily. Another 3-day bladder diary and Overactive Bladder questionnaire (OAB-q) was completed by each subject at the end of a 6-week treatment with Toviaz.
  No washout period.
Groups:
- Fesoterodine: Females with overactive bladder symptoms were given Fesoterodine 4 mg. daily for six weeks.
  Fesoterodine : Fesoterodine 4 mg. tablet by mouth daily for six weeks
Period: Overall Study
Arm/Group | Fesoterodine
Started | 21
Completed | 14
Not Completed | 7
Not completed — Lost to Follow-up | 4
Not completed — Lack of Efficacy | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: The overall number of participants is 21. The 21 participants that took Fesoterodine were the basis for analysis.
Groups:
- Fesoterodine: Overactive bladder subjects took Fesoterodine 4 mg daily for 6 weeks.
Arm/Group | Fesoterodine
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Bladder Diary to Assess Urinary Frequency at Baseline and at End of 6-week Treatment
Description: Overactive bladder subjects filled out a 3-day bladder diary before starting Fesoterodine and another 3-day bladder diary at the end of taking 6 weeks of Fesoterodine. The bladder diary was used to assess urinary frequency. The average number of urinations (frequency) per day over a period of 3 days before the start of medication and at the end of 6 weeks of medication were compared for each subject and then as a group.
Time Frame: Outcome measure was assessed at baseline and at the end of the 6-week treatment
Measure: Mean (Standard Deviation); unit: urinations/day
Groups:
- Fesoterodine: Females with overactive bladder symptoms will be given fesoterodine 4 mg. daily for six weeks.
  fesoterodine : Fesoterodine 4 mg. tablet by mouth daily for six weeks
Arm/Group | Fesoterodine
Number analyzed (Participants) | 14
urinations/day
  Average number of urinations/day after 6 weeks | 12.32 (4.88)
  Average number of urinations/day at baseline | 10.79 (3.64)
Statistical Analysis 1: Comparison: Fesoterodine; Test type: Superiority or Other; p = 0.19, t-test, 2 sided; Mean Difference (Final Values) = 1.53, Standard Deviation 4.88

2. Secondary Outcome: Overactive Bladder Questionnaire (OAB-q) to Assess Bother From Urinary Frequency at Baseline and at 6 Weeks.
Description: Overactive Bladder subjects answered the Overactive Bladder Questionnaire (OAB-q) before starting Fesoterodine and at the end of taking 6 weeks of Fesoterodine. The OAB-q consists of 8 questions asking how bothered subject was in the past 4 weeks. Questions # 1 (Frequent urination during the daytime hours?); #5 (Nighttime urination?) and #6 (Waking up at night because you have to urinate?) are asking about frequency. Choices of answers are: 1 (Not at all); 2 (A little bit); 3 (Somewhat); 4 (Quite a bit); 5 (A great deal) 6 (A very great deal). Multiple responses to the questionnaire were averaged for each participant at baseline and at 6 weeks and then all participants' answers were totaled and averaged at baseline and at 6 weeks.
Time Frame: Outcome measure was assessed at baseline and after the 6 week visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Fesoterodine
Number analyzed (Participants) | 21
scores on a scale
  OAB-q to assess bother from frequency at baseline | 4.89 (0.87)
  OAB-q to assess bother from frequency at 6 weeks | 3.50 (1.45)
Statistical Analysis 1: Comparison: Fesoterodine; Test type: Superiority or Other; p = 0.0021, t-test, 2 sided; Mean Difference (Final Values) = 1.39, Standard Deviation 0.87

3. Primary Outcome: Bladder Diary (Using Urinary Sensation Scale Found in Bladder Diary) to Assess Urinary Urgency at Baseline and at 6-week Treatment
Description: The Urinary Sensation Scale found in the bladder diary given to subjects was used to assess urinary urgency. The Urinary Sensation Scale was filled out by the subject for 3 days before starting Fesoterodine and filled out again for 3 days at the end of taking 6 weeks of Fesoterodine. The scale ranges from 1 (no feeling of urgency), 2 (mild), 3 (moderate), 4 (severe) to 5 (unable to hold; leak urine). The urgency scale with the most check marks per day over a period of 3 days before start of medication was averaged for each subject. The urgency scale with the most check marks per day over a period of 3 days at the end of taking 6 weeks of medication was averaged for each subject. Then, the average before start of medication for all subjects and the average at the end of taking 6 weeks of medication for all subjects were compared.
Time Frame: Outcome measure was assesses at baseline and at the end of the 6-week treatment period.
Measure: Mean (Standard Deviation); unit: scores on Urinary Sensation Scale
Arm/Group | Fesoterodine
Number analyzed (Participants) | 21
scores on Urinary Sensation Scale
  USS to assess baseline urgency | 2.84 (1.02)
  USS to assess 6 week urgency | 2.50 (1.16)
Statistical Analysis 1: Comparison: Fesoterodine; Test type: Superiority or Other; p = 0.18, t-test, 2 sided; Mean Difference (Final Values) = 0.34, Standard Deviation 1.02

4. Secondary Outcome: Overactive Bladder Questionnaire (OAB-q) Will be Used to Assess Bother From Urinary Urgency at Baseline and at 6 Weeks..
Description: Overactive bladder subjects answered the Overactive Bladder questionnaire (OAB-q) before starting Fesoterodine and at the end of taking 6 weeks of Fesoterodine. The OAB-q consists of 8 questions asking how bothered subject was in the past 4 weeks. Questions #2 (An uncomfortable urge to urinate?); #3 (A sudden urge to urinate with little or no warning?); #4 (Accidental loss of small amounts of urine?); #7 (An uncontrollable urge to urinate?); #8 (Urine loss associated with a strong desire to urinate?) are asking about urgency. Choices for answers are: 1 (Not at all); 2 (A little bit); 3 (Somewhat); 4 (Quite a bit); 5 (A great deal); 6 (A very great deal). Multiple responses to the questionnaire was averaged per participant at baseline and at 6 weeks and then all participants answers were totaled and then averaged at baseline and at 6 weeks.
Time Frame: Outcome measures were assessed at baseline and after the 6 week visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Fesoterodine
Number analyzed (Participants) | 21
scores on a scale
  OAB-q to measure bother from urgency at baseline | 4.52 (1.34)
  OAB-q to measure bther from urgency at 6 weeks | 3.14 (1.46)
Statistical Analysis 1: Comparison: Fesoterodine; Test type: Superiority or Other; p = 0.0025, t-test, 2 sided; Mean Difference (Final Values) = 1.38, Standard Deviation 1.34

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at the 6-week follow-up clinic visit. Subjects were also instructed to call if there are any adverse events after the 6-week follow-up visit if they continue on the medication.
Arm/Group | Fesoterodine
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

LIMITATIONS AND CAVEATS:
No serious adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes